CLINICAL TRIAL: NCT05086588
Title: A Prospective, Open-label, Comparative Clinical Study to Evaluate the Safety and Efficacy of BIO-BLUE 90 PLUS With ILM-Blue® as Staining Agent in Vitreo Retinal Surgery.
Brief Title: Safety and Efficacy Evaluation of Two Different Brilliant Blue G Dyes as Staining Agent in Vitreo Retinal Surgery.
Status: Completed | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Aysu Karatay Arsan, Assoc. Prof. MD, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: BTOPL-BBG-001
Record Dates: First submitted 2021-09-24; First posted 2021-10-21 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Macular Holes; Epiretinal Membrane
Keywords: Brilliant Blue G Dye; ILM Pealing; Macular Hole
MeSH Terms: conditions — Retinal Perforations; Epiretinal Membrane

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bio Blue 90 Plus: Patients who were underwent Macular Surgery using Bio Blue 90 Plus (Brilliant Blue G Dye; 0.25 g /l concentration in 0.5 ml BD Glass Syringe; Biotech Vision Care Pvt. Ltd., Ahmedabad, India.)
- ILM Blue: Patients who were underwent Macular Surgery using ILM Blue (Brilliant Blue G Dye; 0.25 g /l concentration in 0.5 ml BD Glass Syringe; D.O.R.C. Dutch Ophthalmic Research Center (International) B.V., Zuidland, The Netherlands)

SUMMARY:
This is a prospective, Open-label, comparative clinical study to asses two brilliant blue G dyes as staining agent in Vitro Retinal Surgery.

DETAILED DESCRIPTION:
The study was designed as prospective, open label, comparative observational study. The patients over 18 years old and undergone Macular Surgery, Internal Limiting membrane removal surgery or vitreomacular traction using the two brilliant blue G dyes as staining agent in Vitro Retinal Surgery were planned to enroll the study. Two blue G dyes (Bio Blue 90 plus and ILM Blue) was randomly assigned at the subject's initial intraoperative visit, according to a computer-generated randomization schedule. During the pars plana vitrectomy, Bio Blue 90 Plus or ILM Blue dyes were injected into eye to stain ILM. Injected Dye was removed from the eye at the end of study before injecting long term tamponade. A total of 5 visits were conducted during the study. Out of them pre-operative visit was done on 1 visit, Surgery/Intraoperative visit and thereafter there were three follow-up visits. The follow- up visits were performed at 1 month, 3 months and 6 Months after the completion of Surgery. Clinical evaluation will be done recording and using staining Ability of ILM (Intra-Operatively), Visualization of Stained Membrane (Intra-Operatively),OCT parameters: (Pre-Op & Post-Op Follow-Up), FFA parameters: (Pre-Op & Post-Op Follow-Up),Fundus auto fluorescence (FAF), Multifocal ERG (Pre-Op & Post-Op Follow-Up) and Visual Field analyses (Pre-Op & Post-Op Follow-Up).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Patient undergone Macular Surgery, Epiretinal membrane removal surgery or vitreomacular traction using the study device
* Patient who can attend all the regular follow-up examinations as per the routine schedule.
* Willingness to adhere to the protocol requirements as evidenced by the informed consent form (ICF) duly read signed and dated by the patient.

Exclusion Criteria:

* Standard exclusion criteria for Macular Surgery like trauma history, previous macular surgery, rhegmatogenous retinal detachment together with macular hole, myopia higher than 10 diopter (D), macular hole for more than 2 years and previous retinal vessel disease.
* Participated in any study during the use of the study device.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were underwent Macular Surgery using study devices were included in the study
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2018-04-04 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Staining Ability of ILM | Intra-Operatively
  Staining of ILM is assed after dye injection with choosing Excellent/Good/ Needs to Improve by surgeon
Change from Baseline to 1 Month, 3 Months and 6 Months in CMT (Central Macular Thickness) | Pre-Op, 1 Month, 3 Month and 6 Month
  CMT (Central Macular Thickness) in micron meters is accessed with ocular coherence tomography
Change from Baseline to 1 Month, 3 Months and 6 Months in TMV ( Total Macular Volume) | Pre-Op, 1 Month, 3 Month and 6 Month
  TMV ( Total Macular Volume) in cubic millimeter is accessed with ocular coherence tomography
Change from Baseline to 1 Month, 3 Months and 6 Months in SFCT (sub foveal choroidal thickness) | Pre-Op, 1 Month, 3 Month and 6 Month
  SFCT (sub foveal choroidal thickness) in cubic meter is accessed with ocular coherence tomography
Change from Baseline to 1 Month, 3 Months and 6 Months in Intra-retinal cuff pathology segmentation | Pre-Op, 1 Month, 3 Month and 6 Month
  Intra-retinal cuff pathology segmentation in micron meter is accessed with ocular coherence tomography
Change from Baseline to 1 Month, 3 Months and 6 Months in RNFL Thickness (Retinal Nerve Fiber Layer) | Pre-Op, 1 Month, 3 Month and 6 Month
  RNFL Thickness (Retinal Nerve Fiber Layer) in micron meter is accessed with ocular coherence tomography
Change from Baseline to 1 Month, 3 Months and 6 Months in Hole diameter | Pre-Op, 1 Month, 3 Month and 6 Month
  Hole diameter in micron meter is accessed with ocular coherence tomography
Change from Baseline to 1 Month, 3 Months and 6 Months in Optic Disc situation | Pre-Op, 1 Month, 3 Month and 6 Month
  Optic Disc situation is accessed with ocular coherence tomography
Change from Baseline to 6 Month in Foveal perfusion characteristics | Pre-Op, 6 Month
  Foveal perfusion characteristics are assed with FFA(Fundus Fluorescein Angiography)
Change from Baseline to 6 Month in Vascular evaluation | Pre-Op, 6 Month
  Vascular evaluation is assed with FFA(Fundus Fluorescein Angiography)
Change from Baseline to 6 Month in Fundus auto fluorescence (FAF) | Pre-Op, 6 Month
  Fundus auto fluorescence (FAF) are assed with FFA(Fundus Fluorescein Angiography)
Multifocal ERG | Pre-op, 1 Month, 3 Month and 6 Month
  During multifocal ERG testing, the patient views a rapidly changing sequence on the monitor. The resulting electrical activity is recorded by an electrode, then amplified and analyzed. During stimulation the hexagons on the screen independently change every 13 milliseconds. They all follow the same pseudorandom sequence, with each hexagon starting at a slightly different position in this sequence. Using a cross-correlation technique, the software determines the retinal response from each of the 103 segments of the retina.
Overview of Adverse Events | Through study completion, an average of 6 Months
  An AE could be any unfavorable and unintended symptom, sign, disease or condition, or test abnormality whether or not considered related to the investigational product. A serious adverse event (SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent AEs (TEAE): AEs that developed/worsened during the 'on treatment period' (from first dose of study device until the end of study period). Category "AE" included participant with both serious and non-serious AE.

SECONDARY OUTCOMES:
Visualization of Stained Membrane | Intra-Operatively
  Visualization of Membrane is assed before and after dye injection with choosing poor/good options by surgeon
Visual Field Analyses | Pre-op, 1 Month, 3 Month and 6 Month
  A test that measures the extent and distribution of the field of vision. A visual field test is done via automated perimetry.
Best Corrected Visual Acuity | Pre-op, 1 Month, 3 Month and 6 Month
  Monocular visual acuity for each eye is be assessed using ETDRS charts held at 4 M.

CONTACTS AND LOCATIONS:
Overall Officials: Aysu Karatay Arsan, MD, Principal Investigator — KARTAL DR. LÜTFİ KIRDAR ŞEHİR HASTANESİ
Locations (1):
- Kartal Dr. Lütfi Kirdar Şehir Hastanesi, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided